CLINICAL TRIAL: NCT05171946
Title: Phase-I, Single Center, Randomized, Dosage Finding Study, to Evaluate the Safety, Tolerability, and Immunogenicity of a Prophylactic COVID-19 pDNA Vaccine After Multiple Ascending Doses in Healthy Adults
Brief Title: Phase-I Study to Evaluate the Safety and Immunogenicity of a Prophylactic pDNA Vaccine Candidate Against COVID-19 in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Iman Almansour (Other)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor-Investigator, Iman Almansour, Clinical Trial Manager, Imam Abdulrahman Bin Faisal University
Organization: Imam Abdulrahman Bin Faisal University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: IAU-1-001-2021
Record Dates: First submitted 2021-12-07; First posted 2021-12-29 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Safety; Vaccine Reaction; Vaccine Adverse Reaction; Immunization; Infection
Keywords: Vaccine; COVID-19; SARS-CoV-2; pDNA vaccine; Phase-I; Prophylactic; Safety; Immunogenicity
MeSH Terms: conditions — Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Low-Dose, 1mg, 3 doses 21 days apart
  Interventions: Drug: S.opt.FL COVID-19 pDNA vaccine
- Cohort 2 (Experimental): Mid-Dose, 2 mg, 2 doses 21 days apart
  Interventions: Drug: S.opt.FL COVID-19 pDNA vaccine
- Cohort 3 (Experimental): High-Dose, 4 mg, 2 doses 21 days apart
  Interventions: Drug: S.opt.FL COVID-19 pDNA vaccine

INTERVENTIONS:
Drug: S.opt.FL COVID-19 pDNA vaccine — Low-Dose: (1mg) level
  Other Names: Almansour-001
  Arms: Cohort 1
Drug: S.opt.FL COVID-19 pDNA vaccine — Mid-Dose: (2mg) level
  Other Names: Almansour-001
  Arms: Cohort 2
Drug: S.opt.FL COVID-19 pDNA vaccine — High-Dose: (4mg) level
  Other Names: Almansour-001
  Arms: Cohort 3

SUMMARY:
A pneumonia of unknown cause detected in Wuhan, China, was first reported in December 2019. On 08 January 2020, the pathogen causing this outbreak was identified as a novel coronavirus 2019. The outbreak was declared a Public Health Emergency of International Concern on 30 January 2020. On 12 February 2020, the virus was officially named as severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), and the WHO officially named the disease caused by SARS-CoV-2 as coronavirus disease 2019 (COVID-19). On 11 March 2020, the WHO upgraded the status of the COVID-19 outbreak from epidemic to pandemic, which is now spreading globally at high speed.

There are currently few licensed vaccines to prevent infection with SARS-CoV-2 or COVID-19 and the duration of response is unknown. Given the rapid transmission of COVID-19 and incidence of disease on a worldwide basis, the rapid development of effective vaccines with sufficient protection and duration of response is of utmost importance.

IAU has developed a thermally stable plasmid DNA (pDNA)-based vaccine candidate using a platform approach that enables the rapid development of vaccines against emerging viral diseases, including SARS-CoV-2. The pDNA vaccine developed by IAU is a synthetic, codon-optimized, encode either the full-length Spike (S) gene or S1 domain of SARS-CoV-2 as genes of interest. Here, we aim to test a synthetic, codon optimized pDNA encoding S.opt.FL as vaccine candidate against COVID-19.

A key advantage of pDNA vaccine is that multiple immunization can be used without the limitations of anti-vector responses.

This study is intended to investigate the safety, immunogenicity, and tolerbilty of this prophylactic vaccine against COVID-19 administered as intramuscular immunization (i.m.).

DETAILED DESCRIPTION:
Sever Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) is a newly emerging coronavirus that is known to cause worldwide public health crisis and an ongoing pandemic since February 2020 with 219 million cases and 4.5 million deaths as of September 2021 (1). The World Health Organization (WHO) has given the term Coronavirus Diseases 19 (COVID-19) to indicate the illness caused by SARS-CoV-2. Individuals infected SARS-CoV-2 can have wide ranges of symptoms that varies between mild to very severe (1,2).

Despite the existence of several COVID-19 vaccine that are approved under emergency use by EMA and FDA (2,3,4,5,6,7), there is a global demand for the manufacturing of sufficient vaccine to control the COVID-19 worldwide. In addition, there is a demand for the development and deployment of new COVID-19 vaccine that is generic and thermally stable for which the vaccine can be stored for a longer period, especially in countries that lacks the infrastructure capabilities to store the vaccine under freezing temperature.

Imam Abdulrahman Bin Faisal University (IAU) has developed an investigational prophylactic COVID-1 pDNA vaccine using a codon optimized spike gene of the SARS-CoV-2 (S.opt.FL). The developed pDNA vaccine possess several advantages; Unlike with mRNA vaccine platforms, pDNA is more stable. Therefore, cold-chain shipment and storage is not needed. Also, the chance for anti-vector immunity generated after immunization viral vector vaccine platform is omitted in pDNA vaccine platform. Importantly, the pDNA can stimulate humoral and cellular immune responses (9,10,11).

IAU COVID-19 vaccine Almansour-001 consists of a plasmid DNA (pDNA) carrying a synthetic, codon-optimized, gene insert that encodes spike (S) gene of COVID-19. The pDNA included in the study is (pVAX-1), an FDA approved plasmid for the application in clinical trials.

Preclinical study conducted at Imam Abdulrahman Bin Faisal University (IAU) have demonstrated that S.opt.FL and S1.opt are immunogenic in mice (8). The study investigated 3 doses versus 4 doses of DNA vaccine. The study demonstrated three doses S1.opt.FL elicited high bAB and nAB responses (8) as well as interferon-Gamma as an indicator of cellular immunity. Previous work on pDNA vaccines encoding the S gene of SARS-CoV, MERS-CoV, and SARS-CoV-2 have demonstrated that pDNA vaccine is safe and well tolerated (12,13,14,15).

The purpose of this clinical trial is to evaluate the safety and immunogenicity of 2 or 3 dose regimen of investigational pDNA vaccine encoding S.opt.FL gene inserted into pVAX1 plasmid (Almansour-001). Here, in this phase-I study, the pDNA vaccine candidate is administered intramuscularly (IM) by immunizing healthy adults (18-55 years). The S.opt.FL pDNA vaccine is evaluated in dose wise manner in three different cohorts (cohort 1: low dosage of pDNA vaccine "1 mg", cohort 2: middle dosage of pDNA vaccine "2 mg", cohort 3: high dosage of pDNA vaccine "4 mg")

ELIGIBILITY:
Inclusion criteria

Study participants should meet ALL the below inclusion criteria to be eligible for the study:

1. Male or female participants between the age of 18 to 55 years (inclusive) at the time of enrollment.
2. Healthy participants as determined by the medical history, physical examination, clinical verification by the investigator.
3. Participant who are committed to comply with planned scheduled visits, vaccination, laboratory tests, and any other procedures.
4. Participants who received 2 doses of an approved mRNA COVID-19 vaccine at least 4 months prior to enrollment.
5. Female subjects must have used an acceptable contraceptive method for at least 60 days prior to receiving the first dose of the investigational vaccine and should continue using contraception for at least 1 month after receiving the last dose of the investigational vaccine.
6. Male subjects able to father children, and sexually active with a female partner who is able to bear children must be willing to use (or have his female partner use) an acceptable contraceptive method from the time they receive the first dose of the study vaccine until at least 1 month after the last dose of study vaccine.
7. Willing to sign the informed consent which includes all the requirements and restrictions listed in the informed consent and the protocol.

Exclusion criteria

Study participants should meet NONE of the exclusion criteria listed below:

1. Participant with known infection with Hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV).
2. Individuals with current infection and diagnosis with COVID-19 documented by PCR nasal swab test.
3. Individuals who received an authorized mRNA COVID-19 vaccine within the past 4 months of first study drug administration.
4. Individuals who received only one dose of a COVID-19 vaccine.
5. Individuals working in facility with high probability of infection with SARS-CoV-2 such as health workers in hospitals.
6. History of adverse reaction associated with vaccines and/or severe allergic reaction to any component of the study intervention.
7. Individuals under immunosuppressive therapy.
8. Individuals receiving treatment or medications that can adherently affect the immune system in the last 90 days, including but not limited to: interferon, immunoglobin, immunomodulators, epinephrine injector, cytotoxic drug.
9. Individuals diagnosed any diseases that is/are associated with sever COVID-19, including the following factors:

   * Diabetes
   * Hypertension
   * Asthma
   * BMI more than 30 kg/m2
   * Pregnant or lactating women.
   * Chronic pulmonary disease
   * Chronic liver diseases
   * Chronic renal diseases
10. Individuals with known or suspected immunological disorders, including, autoimmune disease and diabetes mellitus.
11. Individuals with current or previous neurological disorders, such as seizure or Gillian-Barre syndrome.
12. Individuals with psychiatric disorder or cognitive impairment.
13. Individuals with bleeding disorder or other conditions associated with prolonged bleeding time.
14. Individuals with clinically significant abnormal safety laboratory results at screening in the opinion of the investigator.
15. Individuals receiving or planning to receive non-study vaccine 30 days prior to study enrollment.
16. Individuals receiving or donating blood or blood components 60 days prior to study enrollment.
17. Individuals participating in a clinical trial with an investigational vaccine, treatment, or device 30 days prior to study enrollment.
18. Individuals intending to participate in another clinical trial while being enrolled in this study.
19. Individuals with history of alcohol or drug addiction.
20. Individual with other condition that may interfere with the health or the participants or that interfere with study's primary or secondary objectives.
21. Female participants who are pregnant, plan to get pregnant or are breast feeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
The percentage and frequency of study subjects reporting local reaction | Through 10 days after receiving each dose
The percentage of study subjects reporting systematic reaction | Through 30 days after receiving each dose
The percentage and frequency of study subjects reporting adverse events (AE) | From dose 1 through six months after last dose
The percentage and frequency of study subjects reporting systemic events (SAE) | From dose 1 through six months after last dose
GMT of the serum SARS-CoV-2 binding antibodies (anti-S, anti S1, and anti-RBD) | At baseline (pre-vaccination) and one month after last dose
Proportion of subjects with four folds increase in serum SARS-CoV-2 binding antibodies (anti-S, anti S1, and anti- RBD) | At baseline (pre-vaccination) and one month after last dose
GMT of the serum SARS-CoV-2 S neutralizing antibodies | At baseline (pre-vaccination) and one month after last dose
Proportion of subjects with four folds increase in serum SARS-CoV-2 neutralizing antibodies | At baseline (pre-vaccination) and one month after last dose

SECONDARY OUTCOMES:
GMT of the serum SARS-CoV-2 binding antibodies (anti-S, anti S1, and anti-RBD) | At baseline (pre-vaccination), three weeks after dose 1, three weeks after dose 2, one month after dose 3
Proportion of subjects with four folds increase in serum SARS-CoV-2 binding antibodies (anti-S, anti S1, and anti- RBD) | At baseline (pre-vaccination), three weeks after dose 1, three weeks after dose 2, one month after dose 3
GMT of the serum SARS-CoV-2 neutralizing antibodies | At baseline (pre-vaccination), three weeks after dose 1, three weeks after dose 2, one month after dose 3
Proportion of subjects with four folds increase in serum SARS-CoV-2 neutralizing antibodies | At baseline (pre-vaccination), three weeks after dose 1, three weeks after dose 2, one month after dose 3

OTHER OUTCOMES:
GMT of SARS-CoV-2 S specific binding antibodies against SARS-CoV-2 variants of concern (Alpha, Beta, Gamma, and Omicron) | At baseline (pre-vaccination) and one month after last dose
  V-PLEX SARS-CoV-2 Panel 28 IgG
GMT of SARS-CoV-2 S specific neutralizing antibodies against SARS-CoV-2 variants of concern (Alpha, Beta, Gamma, and Omicron) | At baseline (pre-vaccination) and one month after last dose
  V-PLEX SARS-CoV-2 Panel 28 ACE2
Evaluation of intracellular cytokine responses | At baseline (pre-vaccination), three weeks after dose 1, three weeks after dose 2, one month after dose 3
  Analysis of post-culture PBMCs under 3 conditions with the following panel:IFN-Gamma, TNF, IL-2, IL-4, IL-13 (V-Plex Viral Panel human Kit)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viner RM, Ward JL, Hudson LD, Ashe M, Patel SV, Hargreaves D, Whittaker E. Systematic review of reviews of symptoms and signs of COVID-19 in children and adolescents. Arch Dis Child. 2021 Jul 19;106(8):802-807. doi: 10.1136/archdischild-2020-320972. PMID 33334728
- [Background] Chen X, Laurent S, Onur OA, Kleineberg NN, Fink GR, Schweitzer F, Warnke C. A systematic review of neurological symptoms and complications of COVID-19. J Neurol. 2021 Feb;268(2):392-402. doi: 10.1007/s00415-020-10067-3. Epub 2020 Jul 20. PMID 32691236
- [Background] Oliver SE, Gargano JW, Marin M, Wallace M, Curran KG, Chamberland M, McClung N, Campos-Outcalt D, Morgan RL, Mbaeyi S, Romero JR, Talbot HK, Lee GM, Bell BP, Dooling K. The Advisory Committee on Immunization Practices' Interim Recommendation for Use of Moderna COVID-19 Vaccine - United States, December 2020. MMWR Morb Mortal Wkly Rep. 2021 Jan 1;69(5152):1653-1656. doi: 10.15585/mmwr.mm695152e1. PMID 33382675
- [Background] Oliver SE, Gargano JW, Marin M, Wallace M, Curran KG, Chamberland M, McClung N, Campos-Outcalt D, Morgan RL, Mbaeyi S, Romero JR, Talbot HK, Lee GM, Bell BP, Dooling K. The Advisory Committee on Immunization Practices' Interim Recommendation for Use of Pfizer-BioNTech COVID-19 Vaccine - United States, December 2020. MMWR Morb Mortal Wkly Rep. 2020 Dec 18;69(50):1922-1924. doi: 10.15585/mmwr.mm6950e2. PMID 33332292
- [Background] Roncati L, Roncati M. Emergency use authorization (EUA), conditional marketing authorization (CMA), and the precautionary principle at the time of COVID-19 pandemic. J Public Health Policy. 2021 Sep;42(3):518-521. doi: 10.1057/s41271-021-00299-6. Epub 2021 Jul 27. No abstract available. PMID 34316006
- [Background] MacNeil JR, Su JR, Broder KR, Guh AY, Gargano JW, Wallace M, Hadler SC, Scobie HM, Blain AE, Moulia D, Daley MF, McNally VV, Romero JR, Talbot HK, Lee GM, Bell BP, Oliver SE. Updated Recommendations from the Advisory Committee on Immunization Practices for Use of the Janssen (Johnson & Johnson) COVID-19 Vaccine After Reports of Thrombosis with Thrombocytopenia Syndrome Among Vaccine Recipients - United States, April 2021. MMWR Morb Mortal Wkly Rep. 2021 Apr 30;70(17):651-656. doi: 10.15585/mmwr.mm7017e4. PMID 33914723
- [Background] Krause PR, Gruber MF. Emergency Use Authorization of Covid Vaccines - Safety and Efficacy Follow-up Considerations. N Engl J Med. 2020 Nov 5;383(19):e107. doi: 10.1056/NEJMp2031373. Epub 2020 Oct 16. No abstract available. PMID 33064383
- [Background] Almansour I, Macadato NC, Alshammari T. Immunogenicity of Multiple Doses of pDNA Vaccines against SARS-CoV-2. Pharmaceuticals (Basel). 2021 Jan 6;14(1):39. doi: 10.3390/ph14010039. PMID 33419184
- [Background] Yang B, Jeang J, Yang A, Wu TC, Hung CF. DNA vaccine for cancer immunotherapy. Hum Vaccin Immunother. 2014;10(11):3153-64. doi: 10.4161/21645515.2014.980686. PMID 25625927
- [Background] Liu MA. A Comparison of Plasmid DNA and mRNA as Vaccine Technologies. Vaccines (Basel). 2019 Apr 24;7(2):37. doi: 10.3390/vaccines7020037. PMID 31022829
- [Background] Lee LYY, Izzard L, Hurt AC. A Review of DNA Vaccines Against Influenza. Front Immunol. 2018 Jul 9;9:1568. doi: 10.3389/fimmu.2018.01568. eCollection 2018. PMID 30038621
- [Background] Modjarrad K, Roberts CC, Mills KT, Castellano AR, Paolino K, Muthumani K, Reuschel EL, Robb ML, Racine T, Oh MD, Lamarre C, Zaidi FI, Boyer J, Kudchodkar SB, Jeong M, Darden JM, Park YK, Scott PT, Remigio C, Parikh AP, Wise MC, Patel A, Duperret EK, Kim KY, Choi H, White S, Bagarazzi M, May JM, Kane D, Lee H, Kobinger G, Michael NL, Weiner DB, Thomas SJ, Maslow JN. Safety and immunogenicity of an anti-Middle East respiratory syndrome coronavirus DNA vaccine: a phase 1, open-label, single-arm, dose-escalation trial. Lancet Infect Dis. 2019 Sep;19(9):1013-1022. doi: 10.1016/S1473-3099(19)30266-X. Epub 2019 Jul 24. PMID 31351922
- [Background] Tebas P, Roberts CC, Muthumani K, Reuschel EL, Kudchodkar SB, Zaidi FI, White S, Khan AS, Racine T, Choi H, Boyer J, Park YK, Trottier S, Remigio C, Krieger D, Spruill SE, Bagarazzi M, Kobinger GP, Weiner DB, Maslow JN. Safety and Immunogenicity of an Anti-Zika Virus DNA Vaccine - Preliminary Report. N Engl J Med. 2017 Oct 4:10.1056/NEJMoa1708120. doi: 10.1056/NEJMoa1708120. Online ahead of print. PMID 28976850
- [Background] Tebas P, Kraynyak KA, Patel A, Maslow JN, Morrow MP, Sylvester AJ, Knoblock D, Gillespie E, Amante D, Racine T, McMullan T, Jeong M, Roberts CC, Park YK, Boyer J, Broderick KE, Kobinger GP, Bagarazzi M, Weiner DB, Sardesai NY, White SM. Intradermal SynCon(R) Ebola GP DNA Vaccine Is Temperature Stable and Safely Demonstrates Cellular and Humoral Immunogenicity Advantages in Healthy Volunteers. J Infect Dis. 2019 Jul 2;220(3):400-410. doi: 10.1093/infdis/jiz132. PMID 30891607
- [Background] Muthumani K, Falzarano D, Reuschel EL, Tingey C, Flingai S, Villarreal DO, Wise M, Patel A, Izmirly A, Aljuaid A, Seliga AM, Soule G, Morrow M, Kraynyak KA, Khan AS, Scott DP, Feldmann F, LaCasse R, Meade-White K, Okumura A, Ugen KE, Sardesai NY, Kim JJ, Kobinger G, Feldmann H, Weiner DB. A synthetic consensus anti-spike protein DNA vaccine induces protective immunity against Middle East respiratory syndrome coronavirus in nonhuman primates. Sci Transl Med. 2015 Aug 19;7(301):301ra132. doi: 10.1126/scitranslmed.aac7462. PMID 26290414